CLINICAL TRIAL: NCT01151228
Title: Bedside Ultrasound Assessment of Gastric Content and Volume. Validating a Mathematical Model Using Gastroscopic Examination
Brief Title: Bedside Ultrasound Assessment of Gastric Content and Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 09-0764-BE
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Gastroscopy
Keywords: gastroscopy; ultrasound; stomach volume; patients having gastroscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Zero volume (Placebo Comparator): Patients will not ingest any apple juice prior to the second ultrasound.
  Interventions: Other: Ultrasound examination followed by ingestion of Apple Juice prior to a second ultrasound procedure, followed by gastroscopic suctioning of stomach content.
- 50 mL (Experimental): Patients will ingest 50 mL apple juice prior to the second ultrasound.
  Interventions: Other: Ultrasound examination followed by ingestion of Apple Juice prior to a second ultrasound procedure, followed by gastroscopic suctioning of stomach content.
- 100 mL (Experimental): Patients will ingest 100 mL apple juice prior to the second ultrasound.
  Interventions: Other: Ultrasound examination followed by ingestion of Apple Juice prior to a second ultrasound procedure, followed by gastroscopic suctioning of stomach content.
- 200 mL (Experimental): Patients will ingest 100 mL apple juice prior to the second ultrasound.
  Interventions: Other: Ultrasound examination followed by ingestion of Apple Juice prior to a second ultrasound procedure, followed by gastroscopic suctioning of stomach content.
- 300 mL (Experimental): Patients will ingest 300 mL apple juice prior to the second ultrasound.
  Interventions: Other: Ultrasound examination followed by ingestion of Apple Juice prior to a second ultrasound procedure, followed by gastroscopic suctioning of stomach content.
- 400 mL (Experimental): Patients will ingest 400 mL apple juice prior to the second ultrasound.
  Interventions: Other: Ultrasound examination followed by ingestion of Apple Juice prior to a second ultrasound procedure, followed by gastroscopic suctioning of stomach content.

INTERVENTIONS:
Other: Ultrasound examination followed by ingestion of Apple Juice prior to a second ultrasound procedure, followed by gastroscopic suctioning of stomach content. — Ultrasound scan of the stomach followed by ingestion of 0, 50, 100, 200, 300, or 400 mL of apple juice, followed by second ultrasound scan of the stomach, followed by gastroscopic suctioning of stomach content.

SUMMARY:
Patients undergoing gastroscopy will undergo two pre-procedure ultrasound scans of the stomach, once on arrival in the unit and on an empty stomach and a second time after consumption of a randomized amount of apple juice (0, 50, 100, 200, 300 or 400 mL). Immediately after ingestion and the second ultrasound scan, subjects will have their gastroscopy which will start by suctioning out the apple juice. Measurements of stomach fluid volume conducted by ultrasound will be compared to the actual volume removed during the gastroscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Weight 50-100 kg
* height greater than 150 cm
* ability to provide informed consent

Exclusion Criteria:

* recent upper GI bleed (within 1 month)
* previous lower esophageal or gastric surgery
* not fasted for 8 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Stomach volume | 1 hour
  Fluid volume in the stomach after ingestion of apple juice will be compared between measurements done with ultrasound vs direct suctioning of fluid from the stomach.

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada